CLINICAL TRIAL: NCT07389551
Title: Comparison of Pregabalin Versus Gabapentin as Pre-emptive Analgesic in Patients Undergoing Orthopedic Surgeries Under Spinal Anesthesia
Brief Title: Comparison of Pregabalin Versus Gabapentin as Pre-emptive Analgesic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Usman-QAMC
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Orthopedic Surgery
MeSH Terms: interventions — Gabapentin; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-G (Experimental): Patients were given a single oral dose of gabapentin 300 mg, with 30 ml of water, one hour prior to administration of spinal anesthesia.
  Interventions: Drug: Gabapentin
- Group-P (Experimental): Patients received pregabalin 150 mg as a single oral dose, with 30 ml of water, one hour prior to administration of spinal anesthesia
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Gabapentin — Patients were given a single oral dose of gabapentin 300 mg, with 30 ml of water, one hour prior to administration of spinal anesthesia.
  Arms: Group-G
Drug: Pregabalin — Patients received pregabalin 150 mg as a single oral dose, with 30 ml of water, one hour prior to administration of spinal anesthesia.
  Arms: Group-P

SUMMARY:
There are extensive gaps in the local data considering pregabalin versus gabapentin as pre-emptive analgesics in patients undergoing orthopedic surgeries under spinal anesthesia. Therefore, the current study was planned with the objective of comparing pregabalin versus gabapentin as pre-emptive analgesics in patients undergoing orthopedic surgeries under spinal anesthesia.

DETAILED DESCRIPTION:
Since postoperative pain in orthopedic surgery, whether neuropathic or nociceptive, presents a significant challenge for both surgeons and patients, knowing the more effective gabapentinoid as a pre-emptive analgesic would help clinicians to offer prolonged timing of first rescue analgesia and less opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Either gender
* Aged 20-60 years
* Undergoing lower limb orthopedic surgeries under spinal anesthesia

Exclusion Criteria:

* Patients with a previous history of spine interventions, including surgery or injections (transforaminal, epidural, or facetal) for pain relief
* Patients under any sort of pain modulation therapy, like transcutaneous electrical nerve stimulation
* Patients had a long-term history of any analgesia use
* Those with psychiatric disorders, alcohol/drug dependence, hepatic, renal, cardiac, or pulmonary abnormalities,
* With a history of allergies to gabapentinoids

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Pain severity | 24 hours
  The severity of pain was analyzed on the visual analogue scale (VAS), with a lower score labelling the effectiveness of the treatment.
Analgesia duration | 24 hours
  The duration of analgesia was measured from awakening to the need of rescue analgesia, when a pain score was more than 3 on VAS.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Usman, Principal Investigator — Bahawal Victoria Hospital/Quid-e-Azam Medical College, Bahawalpur; Ambreen Khan, FCPS, Study Director — Bahawal Victoria Hospital/Quid-e-Azam Medical College, Bahawalpur
Locations (1):
- Victoria Hospital/Qaid-e-Azam Medical College, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.